CLINICAL TRIAL: NCT00688597
Title: An Open-Label, Multicenter Study to Evaluate the Safety, Tolerability, Pharmacodynamics, and Pharmacokinetics of Three Dosing Regimens of Oral AT2220 in Patients With Pompe Disease
Brief Title: Study to Evaluate the Safety of AT2220 (Duvoglustat) in Pompe Disease
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Per protocol, 3 sequential dose cohorts were planned. Study discontinued by Sponsor based upon serious adverse events in first 2 of 3 participants in Cohort 1.
Sponsor: Amicus Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: POM-CL-201
Record Dates: First submitted 2008-05-30; First posted 2008-06-03 (Estimated); Results first posted 2018-08-17 (Actual); Last update posted 2025-09-11 (Actual); Status verified 2025-09

CONDITIONS: Pompe Disease
Keywords: Amicus Therapeutics; Duvoglustat; AT2220
MeSH Terms: conditions — Glycogen Storage Disease Type II | interventions — 1-Deoxynojirimycin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Cohort 1 (Experimental): Regimen 1: Low-dose duvoglustat (2.5 grams [g]) once a day (QD) for 3 days, followed by no drug for 4 days, for 11 weeks.
  Interventions: Drug: Duvoglustat
- Cohort 2 (Experimental): Regimen 1: High-dose duvoglustat (5.0 g) QD for 3 days, followed by no drug for 4 days, for 11 weeks.
  Interventions: Drug: Duvoglustat
- Cohort 3 (Experimental): Regimen 2: High-dose duvoglustat (5.0 g) QD for 7 days, followed by no drug for 7 days, for 11 weeks.
  Interventions: Drug: Duvoglustat

INTERVENTIONS:
Drug: Duvoglustat — Powder in a bottle for dissolution in water for oral administration
  Other Names: Duvoglustat hydrochloride; 1-Deoxynojirimycin hydrochloride; AT2220

SUMMARY:
The main purpose of this study was to determine the safety and tolerability of 3 different doses of duvoglustat (AT2220) in participants affected by Pompe disease. The study also evaluated the effects of duvoglustat on functional parameters in Pompe disease.

DETAILED DESCRIPTION:
This was a Phase 2, open-label study in participants with Pompe disease, a lysosomal storage disorder. Duvoglustat is designed to act as a pharmacological chaperone of alpha-glucosidase, in order to restore enzyme activity. This study consisted of a 28-day screening period, an 11-week treatment period, and a 1-week follow-up period. Three dosing regimens of oral duvoglustat were to be evaluated (Cohort 1: 2.5 g daily for 3 days, followed by no study drug for 4 days; Cohort 2: 5 g daily for 3 days, followed by no study drug for 4 days; Cohort 3: 5 g daily for 7 days, followed by no study drug for 7 days).

Participants meeting all eligibility criteria underwent physical examination, electrocardiogram, spirometry, muscular strength test, functional muscle test, 6-minute walk test (when appropriate), laboratory tests, magnetic resonance imaging, and muscle (needle) biopsy. Quality of life was assessed via the 36-Item Short Form Health Survey questionnaire. Functional ability and level of handicap was assessed by Rotterdam handicap scale.

ELIGIBILITY:
Inclusion Criteria:

* Male or female, 18 to 74 years of age inclusive
* Diagnosis of Pompe disease based on clinical assessment, enzyme assay, and/or genotyping. Confirmatory genotyping will be performed on all participants who are screened for the study
* Naïve to enzyme replacement therapy (ERT) or has not received ERT in the 3 months prior to screening
* Willing not to initiate ERT or other prohibited treatment during study participation
* Functional grade for arms and/or legs ≥2 OR sitting forced vital capacity ≥30% and <80% of predicted value, reproducible between screening and baseline (±15%)
* Participants of reproductive potential agree to use reliable methods of contraception during the study
* Participant or legal representative is willing and able to provide written informed consent

Exclusion Criteria:

* Any intercurrent condition that may preclude accurate interpretation of study data
* Obstructive pulmonary disease
* Invasive ventilatory support
* Use of noninvasive ventilatory support >8 hours/day while awake
* History of QTc prolongation >450 milliseconds (msec) for males and >470 msec for females
* History of allergy or sensitivity to the study drug, including any prior serious adverse reaction to iminosugars (such as miglustat or miglitol)
* Pregnancy or breast-feeding
* Current or recent drug or alcohol abuse
* Treatment with another investigational drug within 30 days of study start
* Use of prohibited medications ≤3 months prior to screening
* Otherwise unsuitable for the study in the opinion of the Investigator

Ages: 18 Years to 74 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2008-12-08 (Actual); Primary Completion 2009-12-14 (Actual); Study Completion 2009-12-14 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor Clinical Research, Study Director — Amicus Therapeutics
Locations (1):
- Decatur, Georgia, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3
Started | 3 | 0 | 0
Received at Least 1 Dose of Study Drug | 3 | 0 | 0
Completed | 0 | 0 | 0
Not Completed | 3 | 0 | 0
Not completed — Adverse Event | 2 | 0 | 0
Not completed — Physician Decision | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Safety Population: All participants who received at least 1 dose of duvoglustat.
Groups:
- Cohort 1: Regimen 1: Low-dose duvoglustat (2.5 g) QD for 3 days, followed by no drug for 4 days, for 11 weeks.
- Total: Total of all reporting groups
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3 | Total
Number analyzed (Participants) | 3 | 0 | 0 | 3
Age, Continuous [Mean (Standard Deviation); unit: years] | 49.07 (11.02) |  |  | 49.07 (11.02)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 |  |  | 2
  Male | 1 |  |  | 1

OUTCOME MEASURES:

1. Primary Outcome: Proportion Of Participants Experiencing Severe Treatment-emergent Adverse Events (TEAEs)
Description: The number of participants experiencing severe TEAEs is presented for participants who received duvoglustat treatment in this open-label study. The duration of duvoglustat exposure for Cohort 1 ranged from 2 to 24 days, and their exposure ranged from a total of 7,500 to 32,500 milligrams of duvoglustat. An adverse event (AE) refers to any unfavorable and unintended sign, symptom, syndrome, or illness that develops or worsens during the period of observation in the clinical study. The following guideline was used to grade the intensity of an AE: mild, the AE is easily tolerated and does not interfere with daily activity; moderate, the AE interferes with the daily activity but the participant is still able to function; severe, the AE is incapacitating and requires medical intervention. A summary of serious and all other non-serious AEs regardless of causality is located in the Reported Adverse Events module.
Time Frame: Baseline, Week 11
Population: Safety Population: All participants who received at least 1 dose of duvoglustat.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3
Number analyzed (Participants) | 3 | 0 | 0
Participants | 1 |  |

2. Secondary Outcome: Change In 6-minute Walk Test (6MWT) From Baseline To End Of Study
Description: The 6MWT (American Thoracic Society standards) was evaluated in ambulatory participants at screening, baseline, and to the end of the study. It was a standardized test that measured the distance in meters (m) covered over a 6-minute walk. Reference equations used (for 6MWT distance in healthy adults) included: (height in centimeters [cm], weight in kilograms [kg]) 6MWT distance for men = [7.57 × height (cm)] - [5.02 × age] - [1.76 × weight (kg)] - 309 m; 6MWT distance for women = [2.11 × height (cm)] - [5.78 × age] - [2.29 × weight (kg)] + 667 m
Time Frame: Baseline, Week 11
Population: Safety Population: All participants who received at least 1 dose of duvoglustat.
Measure: Mean (Standard Deviation); unit: m
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3
Number analyzed (Participants) | 3 | 0 | 0
m | -19.660 (41.1845) |  |

ADVERSE EVENTS:
Time Frame: Day 1 (after dosing) through end of follow up.
Description: Due to the discontinuation of the study, AEs were not encoded.
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3
Serious Adverse Events (participants affected / at risk) | 2/3 | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 3/3 | 0/0 | 0/0
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Cohort 1 (N=3) | Cohort 2 (N=0) | Cohort 3 (N=0)
Muscular weakness (General disorders) | 2 | 0 | 0 — [1] The Adverse Event Term was not coded in the database; therefore, "General disorders" was selected as the System Organ Class (SOC) for this AE.
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Cohort 1 (N=3) | Cohort 2 (N=0) | Cohort 3 (N=0)
Muscular weakness (General disorders) | 2 | 0 | 0 — The Adverse Event Term was not coded in the database; therefore, "General disorders" was selected as the SOC for this AE.
Flatulence (General disorders) | 1 | 0 | 0 — The Adverse Event Term was not coded in the database; therefore, "General disorders" was selected as the SOC for this AE.
Abdominal pain upper (General disorders) | 1 | 0 | 0 — The Adverse Event Term was not coded in the database; therefore, "General disorders" was selected as the SOC for this AE.
Alanine aminotransferase increased (General disorders) | 3 | 0 | 0 — The Adverse Event Term was not coded in the database; therefore, "General disorders" was selected as the SOC for this AE.
Aspartate aminotransferase increased (General disorders) | 3 | 0 | 0 — The Adverse Event Term was not coded in the database; therefore, "General disorders" was selected as the SOC for this AE.
Blood creatine phosphokinase increased (General disorders) | 3 | 0 | 0 — The Adverse Event Term was not coded in the database; therefore, "General disorders" was selected as the SOC for this AE.
Fall (General disorders) | 2 | 0 | 0 — The Adverse Event Term was not coded in the database; therefore, "General disorders" was selected as the SOC for this AE.
Dysphagia (General disorders) | 1 | 0 | 0 — The Adverse Event Term was not coded in the database; therefore, "General disorders" was selected as the SOC for this AE.
Joint injury (General disorders) | 1 | 0 | 0 — The Adverse Event Term was not coded in the database; therefore, "General disorders" was selected as the SOC for this AE.

LIMITATIONS AND CAVEATS:
The serious adverse event of muscle weakness was the main contributor to the study not reaching the target number of participants needed to achieve target power and statistically reliable results.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The investigator can only publish the results from this trial provided they supply the sponsor (or authorized entity) a copy of any proposed publication for review. If requested, the investigator will remove information deemed confidential or proprietary by the sponsor and will withhold publication for an additional period of time to allow the sponsor to take appropriate measures to establish and preserve its proprietary rights.